CLINICAL TRIAL: NCT04584983
Title: Bilirubin Neurotoxicity (BN) and Neurodevelopmental Impairment (NDI) in Extremely Preterm (EP) Infants: Avoidable by Reducing the Usual Intravenous Lipid (UL) Administration
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Lindsay Fleig Holzapfel, MD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-0916; KL2TR003168 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bilirubin Encephalopathy
Keywords: preterm; bilirubin; lipid emulsions; unbound bilirubin; unbound free fatty acids
MeSH Terms: conditions — Kernicterus; Premature Birth | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual prescribed intralipid (UL) regimen (Active Comparator)
  Interventions: Drug: usual prescribed intralipid (UL) regimen
- restricted prescribed intralipid (RL) regimen (Experimental)
  Interventions: Drug: restricted prescribed intralipid (RL) regimen

INTERVENTIONS:
Drug: usual prescribed intralipid (UL) regimen — Intralipid will be started at 1 g/kg/day and routinely advanced by 1 g/kg/day each day to a max of 3 g/kg/day as per usual clinical practice
  Arms: usual prescribed intralipid (UL) regimen
Drug: restricted prescribed intralipid (RL) regimen — Intralipid will be started at 0.5 g/kg/day and routinely advanced by 0.5 g/kg/day each day to a max of 1.5 g/kg/day (half rate of usual clinical practice).
  Arms: restricted prescribed intralipid (RL) regimen

SUMMARY:
The purpose of this study is to evaluate the effect of usual versus reduced lipid intake on unbound bilirubin levels, brainstem auditory evoked responses, and neurodevelopmental outcome at 2 years in extremely preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* no major congenital anomaly or overt nonbacterial infection
* mother has consented to inclusion of the infant for the Neonatal Research Network (NRN) Cycled Phototherapy Trial

Exclusion Criteria:

* has received Intralipid

Max Age: 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2026-06-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay F Holzapfel, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holzapfel LF, Arnold C, Tyson JE, Shapiro SM, Reynolds EW, Pedroza C, Stephens EK, Kleinfeld A, Huber AH, Rysavy MA, Del Mar Romero Lopez M, Khan AM. Effect of reduced versus usual lipid emulsion dosing on bilirubin neurotoxicity and neurodevelopmental impairment in extremely preterm infants: study protocol for a randomized controlled trial. BMC Pediatr. 2023 Jul 10;23(1):347. doi: 10.1186/s12887-023-04149-0. PMID 37430233
- [Derived] Holzapfel L, Arnold C, Tyson J, Shapiro S, Reynolds E, Pedroza C, Stephens E, Kleinfeld A, Huber A, Rysavy M, Khan A, Del Mar Romero Lopez M. Effect of Reduced Versus Usual Lipid Emulsion Dosing on Bilirubin Neurotoxicity and Neurodevelopmental Impairment in Extremely Preterm Infants: Study Protocol for a Randomized Controlled Trial. Res Sq [Preprint]. 2023 Mar 7:rs.3.rs-2566352. doi: 10.21203/rs.3.rs-2566352/v1. PMID 36945475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Started | 67 | 67
Received Intervention | 65 | 67
Completed | 65 | 67
Not Completed | 2 | 0
Not completed — Parental request for withdraw | 2 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants who received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Customized [Count of Participants; unit: Participants]
  < 27 weeks gestational age | 62 | 64 | 126
  ≥ 27 weeks gestational age | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 40 | 37 | 77
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 20 | 45
  White | 35 | 37 | 72
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 9 | 11
Region of Enrollment [Number; unit: participants]
  United States | 65 | 67 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Unbound Bilirubin (UB) Concentration Greater Than 30 Nanomoles Per Liter (Nmol/L)
Time Frame: within first 14 days of life
Population: Data were not collected for 8 participants in the usual prescribed intralipid (UL regimen) arm because 1 died before sampling began, and 7 did not receive sampling because they never achieved the maximum dose of lipid and therefore did not trigger blood draws to begin. Data were not collected for 4 participants in the reduced prescribed intralipid (RL) regimen arm because 3 died before sampling began, and 1 did not achieve the maximum dose of lipid and therefore, did not trigger blood draws.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
Participants | 2 | 3

2. Primary Outcome: Average Unbound Bilirubin (UB) Concentration
Description: 6 UB measurements will be taken per participant .Average of the 6 readings will be reported
Time Frame: within first 14 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
nanomolar (nM) | 12.3 (7.8) | 13.2 (7.8)

3. Primary Outcome: Brain Stem Auditory-evoked Response (BAER) V Latency
Description: Brainstem auditory evoked response (BAER) testing is a procedure used to assess the auditory pathways of the brainstem and evaluate hearing ability. Wave latency, measured in milliseconds, is the measure of electric transmission of sound. If the wave latency is prolonged, this means that something is in the way of electric sound wave transmission, such as bilirubin which has an affinity for depositing in a specific area of the brainstem that wave V measures.
Time Frame: 38 weeks post menstrual age(PMA)
Population: Data were not collected from 7 participants in the usual prescribed intralipid (UL regimen) arm who received intervention because 7 infants died in the UL arm before BAER testing was performed at 36 weeks PMA . Data were not collected from 10 participants in the reduced prescribed intralipid (RL) regimen arm because 10 infants died in the UL arm before BAER testing was performed at 36 weeks PMA.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 58 | 57
milliseconds (ms) | 7.25 (0.58) | 7.34 (0.48)

4. Secondary Outcome: Peak Free Fatty Acid Uptake (FFAU)
Time Frame: within first 14 days of life
Population: Data were not collected for 9 participants in the usual prescribed intralipid (UL) regimen arm because 1 died before sampling, 7 didn't receive blood draws because they never achieved the maximum dose of lipid, and 1 didn't have enough serum for testing. Data were not collected for 5 participants in the reduced prescribed intralipid (RL) regimen arm because 3 died before sampling, 1 didn't achieve the maximum dose of lipid for blood draws and 1 didn't have enough serum for testing.
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 56 | 62
nanomolar (nM) | 105.53 (92.76) | 64.39 (81.84)

5. Secondary Outcome: Peak UB Concentration
Time Frame: within first 14 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
nanomolar (nM) | 23.4 (17.5) | 22.0 (17.7)

6. Secondary Outcome: Total Unbound Free Fatty Acids (FFA)
Description: 6 FFA measurements will be taken for each participant.Average of the 6 readings will be reported
Time Frame: within first 14 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
nanomolar (nM) | 41.4 (27.6) | 31.0 (34.2)

7. Secondary Outcome: Peak Total Serum Bilirubin
Time Frame: within first 14 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
milligrams per decilitre (mg/dL) | 5 (1.8) | 5.2 (1.3)

8. Secondary Outcome: Number of Patients With Direct Bilirubin Greater Than 1.5 mg/dL
Time Frame: Before discharge (discharge is on average 3 months after birth)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 57 | 63
Participants | 9 | 10

9. Secondary Outcome: Amount of Protein Given to Participant in Grams Per Kilograms on Day 14 of Life
Description: Calculated as the mean daily protein intake in grams per kilogram of body weight on Day 14 of life.
Time Frame: Day 14 of life
Population: Data were not collected for 7 participants in the usual prescribed intralipid (UL) regimen arm because 6 participants passed away and 1 participant only received carbohydrates therefore the 1 participant did not receive proteins at day 14 of life. Data were not collected for 6 participants in the restricted prescribed intralipid (RL) regimen arm because 6 participants passed away.
Measure: Mean (Standard Deviation); unit: grams per kilograms
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 58 | 61
grams per kilograms | 3.62 (0.56) | 3.60 (0.48)

10. Secondary Outcome: Amount of Carbohydrates Given to Participant in Grams Per Kilograms on Day 14 of Life
Description: Calculated as the mean daily carbohydrates intake in grams per kilogram of body weight on Day 14 of life.
Time Frame: Day 14 of life
Population: Data were not collected for 6 participants in the usual prescribed intralipid (UL) regimen arm because 6 participants passed away. Data were not collected for 6 participants in the restricted prescribed intralipid (RL) regimen arm because 6 participants passed away.
Measure: Mean (Standard Deviation); unit: Grams Per Kilograms
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 59 | 61
Grams Per Kilograms | 13.46 (3.53) | 13.50 (2.74)

11. Secondary Outcome: Amount of Fats Given to Participant in Grams Per Kilograms on Day 14 of Life
Description: Calculated as the mean daily fats intake in grams per kilogram of body weight on Day 14 of life.
Time Frame: Day 14 of Life
Population: Data were not collected for 7 participants in the usual prescribed intralipid (UL) regimen arm because 6 participants passed away and 1 participant only received carbohydrates therefore the 1 participant did not receive fats on day 14 of life. Data were not collected for 6 participants in the restricted prescribed intralipid (RL) regimen arm because 6 participants passed away.
Measure: Mean (Standard Deviation); unit: Grams Per Kilograms
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 58 | 61
Grams Per Kilograms | 4.05 (1.39) | 3.74 (1.68)

12. Secondary Outcome: Weight z Score
Description: Weight Z-scores were calculated using the PediTools Fenton Growth Curves Calculator (2013 version), based on the Fenton Preterm Growth Charts.
  The following thresholds were used for interpretation:
  Z-score ≤ -2: Growth failure (worse outcome)
  Z-score = 0: Population mean (appropriate outcome)
  Z-score 0 to <2: Appropriate growth (better outcome)
  Z-score ≥ 2: Excessive growth (worse outcome)
Time Frame: day 28
Population: Data were not collected for 6 participants in the usual prescribed intralipid (UL) regimen arm because 6 participants passed away. Data were not collected for 7 participants in the restricted prescribed intralipid (RL) regimen arm because 7 participants passed away.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 59 | 60
z-score | -1.019 (0.87) | -0.870 (0.72)

13. Secondary Outcome: Weight
Time Frame: birth
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 65 | 67
grams | 680 [570 to 840] | 700 [610 to 838]

14. Secondary Outcome: Weight
Time Frame: 36 weeks postmenstrual age
Population: Data were not collected from 10 participants in the usual prescribed intralipid (UL) regimen arm because 7 participants passed away and 3 were discharged before 36 weeks. Data were not collected from 14 participants in the restricted prescribed intralipid (RL) regimen arm because 10 participants passed away and 4 were discharged before 36 weeks.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 55 | 53
grams | 1995 (383) | 2077 (300)

15. Secondary Outcome: Number of Patients With Bronchopulmonary Dysplasia
Time Frame: 36 weeks post menstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 65 | 67
Participants | 48 | 55

16. Secondary Outcome: Number of Patients With Perinatal and Hospital Acquired Sepsis Episodes
Time Frame: birth until discharge ( discharge will be about 3 months post birth)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 65 | 67
Participants | 22 | 16

17. Secondary Outcome: Number of Patients Who Died
Time Frame: 24 months PMA
Reporting Status: Not Posted

18. Secondary Outcome: Number of Patients With Neurodevelopmental Impairment
Time Frame: 24 months PMA
Reporting Status: Not Posted

19. Secondary Outcome: Number of Patients With Hearing Loss
Time Frame: 24 months PMA
Reporting Status: Not Posted

20. Secondary Outcome: Number of Patients With Cerebral Palsy
Time Frame: 24 months PMA
Reporting Status: Not Posted

21. Secondary Outcome: Serial FiO2 (Fraction of Inspired Oxygen)
Time Frame: Day 1 of life through day 14 of life
Population: This outcome measure was pre-specified in the protocol; however, no data were collected for this measure. Due to resource limitations, the study team was unable to obtain the required data. Specifically, staffing limitations led to the decision to not collect any data from any participants for this Outcome Measure. Data collection and analysis for this outcome measure will not be conducted in the future. Therefore, no participants were measured or analyzed for this outcome measure.
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Ventilator Setting
Time Frame: Day 1 of life through day 14 of life
Population: as for outcome 21
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 26 months
Arm/Group | Usual Prescribed Intralipid (UL) Regimen | Restricted Prescribed Intralipid (RL) Regimen
All-Cause Mortality (participants affected / at risk) | 7/67 | 10/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04584983/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04584983/ICF_001.pdf